CLINICAL TRIAL: NCT00005739
Title: Behavioral Interventions for Control of Tuberculosis
Brief Title: Behavioral Interventions for Control of TB
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CUMC ID unknown (4948); R01HL055751 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Lung Diseases; Tuberculosis
MeSH Terms: conditions — Lung Diseases; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Community-based therapy (case): Community-based directly observed therapy (DOT) - A community-based intervention conducted by trained graduates of a TB directly observed therapy (DOT) program (peer workers)
  Interventions: Behavioral: Community-based directly observed therapy (DOT)
- Self-administered treatment (control): Clinic directly observed therapy (DOT) - Traditional self-administered preventive treatment
  Interventions: Behavioral: Clinic directly observed therapy (DOT)

INTERVENTIONS:
Behavioral: Community-based directly observed therapy (DOT) — A community-based intervention conducted by trained graduates of a TB directly observed therapy (DOT) program (peer workers)
  Other Names: Community-based DOT
  Groups: Community-based therapy (case)
Behavioral: Clinic directly observed therapy (DOT) — A traditional self-administered preventive treatment
  Other Names: Clinic DOT
  Groups: Self-administered treatment (control)

SUMMARY:
To compare alternative methods to ensure completion of treatment and preventive therapy for tuberculosis (TB) in inner cities, and to identify the most cost-effective methods to accomplish that. The basis for comparison included adherence rates and cost savings as primary outcomes, and other parameters such as patient satisfaction, development of social networks, and participation in support programs as secondary outcomes.

Two clinical trials were conducted with patients from Harlem. Among those with active disease, a clinic-based surrogate family model was compared to traditional community-based directly observed therapy (DOT). Among those eligible for preventive therapy, a community-based intervention conducted by trained graduates of a TB DOT program (peer workers) was compared to traditional self-administered preventive treatment.

DETAILED DESCRIPTION:
Tuberculosis was on the decline from the mid 1950s until the mid 1980s; however, the United States is now experiencing a resurgence of tuberculosis. In 1992, approximately 27,000 new cases were reported, an increase of about 20 percent from 1985 to 1992. Not only are tuberculosis cases on the increase, but a serious aspect of the problem is the recent occurence of outbreaks of multidrug resistant (MDR) tuberculosis, which poses an urgent public health problem and requires rapid intervention.

Control programs involve two major components. First, and of highest priority, is to detect persons with active tuberculosis and treat them with effective antituberculosis drugs, which prevents death from tuberculosis and stops the transmission of infection to other persons. Treatment of active tuberculosis involves taking multiple antituberculosis drugs daily or several times weekly for at least six months. Failure to take the medications for the full treatment period may mean that the disease is not cured and may recur. If sufficient medications are not prescribed early and taken regularly, the tuberculosis organism can become resistant to the drugs, and the drug resistant tuberculosis then may be transmitted to other persons. Drug resistant disease is difficult and expensive to treat, and in some cases, cannot be treated with available medications.

The second major goal of control efforts is the detection and treatment of persons who do not have active tuberculosis, but who have latent tuberculosis infection. These people may be at high risk of developing active tuberculosis. The only approved treatment modality for preventive therapy requires treatment daily or twice weekly for a minimum of six months, and many patients do not complete the full course of therapy. Public and patient programs are needed to increase the awareness of the problems associated with tuberculosis control.

The study is part of the NHLBI initiative "Behavioral Interventions for Control of Tuberculosis" . The concept for the initiative originated from the National Institutes of Health Working Group on Health and Behavior. The Request for Applications was released in October, 1994.

ELIGIBILITY:
Inclusion Criteria:

-Patients with suspected and confirmed TB

Exclusion Criteria:

-Patients that are not a part of the therapy program established at Harlem Hospital, New York City

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected and confirmed TB
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 1995-09; Primary Completion 2004-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visit adherence rate | At the end of study
  Prevalence of suspected and confirmed tuberculosis patients that continued treatment

SECONDARY OUTCOMES:
Treatment completion rate | At end of study
  Prevalence of suspected and confirmed tuberculosis patients that completed treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, Principal Investigator — University Professor; Director, ICAP, Department of Epidemiology
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- Available data/document: Abstract — http://ajph.aphapublications.org/doi/pdf/10.2105/AJPH.86.8_Pt_1.1146